CLINICAL TRIAL: NCT01070719
Title: Pharmacokinetic, Immunological and Biochemical Sample Collection and Analysis of a Tysabri Patient Cohort
Status: Completed | Type: Observational
Sponsor: John F. Foley, MD (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor-Investigator, John F. Foley, MD, Sponsor-Investigator, Rocky Mountain MS Research Group, LLC
Organization: Rocky Mountain MS Research Group, LLC (Other)
Other Study IDs: 001-001-TY
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Multiple Sclerosis; Relapse
Keywords: Multiple Sclerosis, relapsing forms
MeSH Terms: conditions — Multiple Sclerosis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum will be collected, and spun for specific tests. The back-up specimens (plasma)will be held in case of a laboratory error.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Relapsing form of MS treated with natalizumab: Only patients diagnosed with a relapsing form of Multiple Sclerosis (MS) and who are being treated with Tysabri (natalizumab) will be included in this Phase IV observational study.

SUMMARY:
This is an open-label study of patients with relapsing forms of Multiple Sclerosis designed to assess the biochemical, immunological and pharmacokinetic profiles of a large, actively infusing natalizumab patient population. A duration effect for progressive multifocal leukoencephalopathy (PML) risk associated with natalizumab therapy appears to exist. There is minimal data available to understand this effect at the biochemical and cellular level. The purpose of this study is to gather preliminary data on several parameters to guide in more focused research on the duration effect.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Aged 18 to 75 years old, inclusive, at the time of informed consent.
3. Must be a patient with a relapsing form of Multiple Sclerosis enrolled in the TOUCH Prescribing Program who is not expected to discontinue Tysabri® therapy prior to completion of the requirements of this study.
4. Must have been treated with monthly IV infusions of Tysabri® 300 mg for at least 1 month.
5. Must have a magnetic resonance imaging (MRI) brain scan, performed prior to the initiation of treatment with Tysabri®, on file.
6. Must weigh between 42 and 126 kg, inclusive.
7. Fifteen patients who are 1 month to-12 months of natalizumab therapy, fifteen patients who are 24 months and over of natalizumab therapy will be asked to participate in the TNF alpha subset.

Exclusion Criteria:

Medical History:

1. History of, or abnormal laboratory results indicative of, any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.
2. If subject answers 'Yes" to any question on the PML questionnaire that is not resolved prior to infusion as per standard operating procedure for natalizumab infusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsing forms of MS currently being treated with natalizumab.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Foley, MD, Principal Investigator — Rocky Mountain MS Research Group, LLC
Locations (1):
- Rocky Mountain Multiple Sclerosis Clinic, Salt Lake City, Utah, United States